CLINICAL TRIAL: NCT01236820
Title: L5 as a Risk Factor of Cardiovascular Disease in Chronic Kidney Disease and Dialysis Patients
Brief Title: A Study Using L5 as a Risk Factor of Cardiovascular (CV) Disease in Chronic Renal and Dialytic Patients
Acronym: L5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chiu-Ching Huang, China Medical University Hospital
Other Study IDs: CTCHANG001
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Cardiovascular Disease; Chronic Kidney Disease Patients; Hemodialytic Patients; High LDL Level; High L5 Level
Keywords: L5; LDL; Cardiovascular disease; Chronic kidney disease; Hemodialysis
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: Healthy population
- CKD Patients: Chronic Kidney Disease, in Stage III-V
- HD patients: End-stage renal disease patients undergoing hemodialysis

SUMMARY:
The purpose of this study is to determine whether L5, one of the Low Density Lipoproteins, is an effective predicting factor for cardiovascular disease in chronic renal and hemodialytic patients.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the most important cause of death of chronic kidney disease (CKD) and hemodialysis (HD) patients. Low Density Lipoprotein (LDL) is an essential indicator of CVD.The higher the plasma LDL level, the higher the risk of CVD. LDL is a heterogenous substance composed of different mass and size. Oxidized LDL (oxLDL) is the oxidation product of LDL and is the most important component of LDL associated with CVD. The oxLDL is mostly trapped within tissue and not easily to be detected from blood. L5 iw a kind of electronegative LDL and is associated with CVD in smokers and diabetic patients, even if these patients have normal plasma LDL. Uremia patients have lipid profile different from that of general people,while HD Patients have lower LDL and CKD patients have LDL higher than that of general population. Thus LDL plasma level cannot fully explain the high risk of CVD in CKD and HD patients. As patients with normal LDL but high L5 are prone to have CVD, we suspect there might be association of L5 with CVD in both CKD and HD patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of CKD
* clinical diagnosis of HD

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents in Taiwan, mostly in Taichung area
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan